CLINICAL TRIAL: NCT00448773
Title: Effectiveness of Selected Non-pharmaceutical Interventions in Reducing Influenza-like Illness Among University Students
Brief Title: REDucing Influenza Among University Students, University of California at Berkeley
Acronym: REDI-US
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Dr. Tomas Aragon, University of California at Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-20061243
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Influenza-like Illness; Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Behavioral: Online education

SUMMARY:
We will be testing the hypothesis whether online education for UC Berkeley students on respiratory hygiene, cough etiquette, hand hygiene/awareness, as well as face mask use (while ill) will reduce the acquisition and transmission of influenza-like illness. The study will be conducted during the flu seasons 2006-7 and 2007-8.

ELIGIBILITY:
Inclusion Criteria:

* Registered students
* Attending UC Berkeley at least half-time during the study period

Exclusion Criteria:

* Enrolled but studying remotely or abroad for all or part of the study period
* Persons less than 17 years of age

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of influenza-like illness

CONTACTS AND LOCATIONS:
Overall Officials: Tomas J Aragon, MD, DrPH, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States